CLINICAL TRIAL: NCT01787539
Title: The Role of Postoperative Chemotherapy Cycles in the Combined Modality Therapy of Gastric Cancer With Perioperative Chemotherapy and Surgery in Pathological Responders
Brief Title: The Role of Postoperative Cycles in the Perioperative Chemotherapy for Gastric Cancer
Acronym: STOPEROPCHEM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Collaborators: St Johns' Oncology Center in Lublin (Unknown)
Responsible Party: Principal Investigator, Tomasz Skoczylas, MD, PhD, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-COMB-0254/275/2012-MUL; GC-0254/282/2011/275/2012-MUL (Other: Medical University of Lublin)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; perioperative chemotherapy; combined modality therapy; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete Perioperative Chemotherapy (Experimental): Preoperative chemotherapy with EOX regimen: Epirubicin with intravenous bolus at a dose of 50 mg/m2 an on day 1; Oxaliplatin with intravenous infusion during a 2-hour period at a dose of 130 mg/m2; Capecitabine administrated orally at a twice daily dose of 625 mg /m2 during 21 days. Treatment cycles will be repeated every 3 weeks.
  Surgery: total or subtotal gastrectomy with D2 lymph node dissection. The surgical resection will be conducted 4-6 weeks after preoperative chemotherapy.
  Postoperative chemotherapy will be administrated in patients with tumor regression grade 0, 1, 2 randomized to perioperative chemotherapy and will be initiated 6 to 12 weeks after surgery with the same regimen as in the preoperative part.
  Interventions: Drug: Postoperative Chemotherapy
- Preoperative Chemotherapy (No Intervention): Preoperative chemotherapy with EOX regimen: Epirubicin with intravenous bolus at a dose of 50 mg/m2 an on day 1; Oxaliplatin with intravenous infusion during a 2-hour period at a dose of 130 mg/m2; Capecitabine administrated orally at a twice daily dose of 625 mg /m2 during 21 days. Treatment cycles will be repeated every 3 weeks.
  Surgery: total or subtotal gastrectomy with D2 lymph node dissection. The surgical resection will be conducted 4-6 weeks after preoperative chemotherapy.
  Patients with tumor regression grade 0, 1, 2 randomized to preoperative chemotherapy will not undergo postoperative chemotherapy and will be followed-up.

INTERVENTIONS:
Drug: Postoperative Chemotherapy — Postoperative chemotherapy with EOX regimen: Epirubicin with intravenous bolus at a dose of 50 mg/m2 an on day 1; Oxaliplatin with intravenous infusion during a 2-hour period at a dose of 130 mg/m2; Capecitabine administrated orally at a twice daily dose of 625 mg /m2 during 21 days. Treatment cycles will be repeated every 3 weeks.
  Postoperative chemotherapy will be administrated in patients with tumor regression grade 0, 1, 2 randomized to perioperative chemotherapy and will be initiated 6 to 12 weeks after surgery.
  Arms: Complete Perioperative Chemotherapy

SUMMARY:
Taking into account the substantial doubts concerning the potential benefit of postoperative part in the perioperative chemotherapy regimen we designed a study assessing value of this approach in gastric cancer. To improve compliance with a protocol regimen of this aggressive combined therapy we replaced tested in the MAGIC trial ECF regimen with more effective and better tolerable EOX chemotherapy regimen. The value of postoperative three-cycle EOX regimen will be tested in patients with locoregionally advanced gastric cancer with positive pathological response to preoperative three-cycle EOX chemotherapy regimen. The patients will be randomized to the postoperative chemotherapy or to the follow-up arm.

DETAILED DESCRIPTION:
The MAGIC trial, also considered the "milestone" study, definitely proved that neoadjuvant chemotherapy improves the outcome of patients with locally advanced gastric cancer. Resection was considered curative in 79% under combination therapy versus in 69% of only operated patients (P = 0.02), 2-year survival rates were 50 and 41%, and 5-year-survival rates were 36 and 23% (P = 0.009), respectively. The substantial weak point of the MAGIC trial remains the fact that only about 40% of the patients received the full dosage of scheduled postoperative chemotherapy, mainly due to intolerance or toxicity reasons.

The noninferiority in relation to survival of capecitabine to 5-FU in triplet regimens for the treatment of patients with advanced esophagogastric cancer was demonstrated in the large multicenter randomized phase III, REAL-2 study, including 1002 patients. Capecitabine has overcome the doubts concerning the potential efficacy of oral drug administration in patients with gastric carcinoma, especially in relation to those patients who have undergone partial or total gastrectomy. The same study demonstrated the noninferiority of oxaliplatin versus cisplatin in advanced gastric cancer and confirmed the acceptable tolerability profile of this third-generation platinum analogue. It was anticipated that the use of these newer agents as components of triplet regimens would reduce toxicity and thereby render an alternative to the standard ECF combination easier to handle as a consequence of replacing the cisplatin component with oxaliplatin, replacing the infusional 5-fluorouracil component with oral capecitabine in EOX regimen. Furthermore, achieving a median overall survival time of 11.2 months, the EOX regimen appeared to be more active than ECF (median overall survival time, 9.9 months), with the higher 1-year survival rate 47% vs 38%, respectively. Compared with the ECF regimen, EOX was associated with significantly lower rates of grade 3 or 4 neutropenia and grade 2 alopecia, but significantly higher rates of grade 3 or 4 lethargy, diarrhea, and peripheral neuropathy. Based on the results of the REAL study, EOX is therefore tolerable, and at least as active as ECF. This modified regimen could therefore be considered to be a new standard treatment and may be an appropriate reference regimen for future studies in advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed gastric cancer
* potentially resectable, local or locoregional cancer with clinical staging cT2-4aN0-3M0. A clinical assessment of location, resectability and staging will be performed based on endoscopy, barium swallow, endoscopic ultrasound, multidetector computed tomography and diagnostic laparoscopy with cytology washing.
* medically fit to undergo a major abdominal surgery and in general condition allowing to tolerate long-lasting chemotherapy (Karnofsky Performance Status ≥70, ECOG 0-1)

Exclusion Criteria:

* Pregnancy or breast feeding.
* Diagnosed other malignancy and/or chemotherapy administrated within the last 5 years
* Gastric remnant cancer;
* Early Gastric Cancer;
* Irresectable or disseminated cancer with distant organ metastases and/or peritoneal spreading and/or positive cytology washing
* Poor performance status measured by Karnofsky index < 60 or ECOG < 1
* Clinically important active systemic disease: unstable diabetes, circulatory failure of NYHA III or IV, unstable arterial hypertension, unstable coronary heart disease, recent heart infarct or brain insult within the last 6 months, severe COPD, peripheral neuropathy of grade 2-4;
* Severe hematological abnormalities: HGB < 10.0 gm/dL and/or neutropenia < 1500 /mm3; PLT < 100 000 /mm3.
* Severe renal dysfunction requiring peritoneal dialysis, hemodialysis or hemofiltration or oliguria <20ml/h.
* Severe liver dysfunction: acute or chronic hepatitis, liver cirrhosis, liver failure, abnormal liver testing: ALAT or ASPAT or ALP >2.5 - 5.0 × upper limit; total bilirubin >2 x upper limit.
* Concommitant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
cancer free and overall survival | 5 years

SECONDARY OUTCOMES:
overall and severe toxicity rate | 8 weeks
chemotherapy related mortality | 8 weeks
the rate of dose reduction for chemotherapeutics | 3 months
the rate of chemotherapy cessation | 3 months

OTHER OUTCOMES:
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skoczylas, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Grzegorz Wallner, Professor, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Elżbieta Starosławska, MD, PhD, Principal Investigator — St Johns' Oncology Center in Lublin; Tomasz Kubiatowski, MD, PhD, Principal Investigator — St Johns' Oncology Center in Lublin
Locations (2):
- Poland (2):
  - Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin, Lublin, Lublin Voivodeship
  - St. John's Cancer Center, Lublin, Lublin Voivodeship